CLINICAL TRIAL: NCT01671085
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3015014 in Subjects With Elevated LDL-C on a Stable Statin Therapy
Brief Title: A Study of LY3015014 in Healthy Participants With High Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14938; I5S-EW-EFJD (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — frovocimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 milligrams per kilogram (mg/kg) of LY3015014 (Experimental): 1.0 mg/kg of LY3015014 given subcutaneously (SQ) on 2 dosing occasions occurring 4 weeks apart (Q4W) (Days 1 and 29).
  Interventions: Drug: LY3015014
- Placebo (Placebo Comparator): 0.9% sodium chloride injection given SQ (to match LY3015014) on 2 dosing occasions Q4W (Days 1 and 29).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3015014 — Administered SQ
  Arms: 1.0 milligrams per kilogram (mg/kg) of LY3015014
Drug: Placebo — Administered SQ
  Arms: Placebo

SUMMARY:
This is a study in healthy participants with high levels of "bad" cholesterol who are already taking a popular type of cholesterol-lowering medication called statins. Following multiple doses of LY3015014, investigators will study the safety and tolerability of the drug, how the body handles the drug, and the drug's effect on the body. Participants will remain in the study for about 3 months, not including screening. Screening is required within 28 days before the study starts.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy males or females without childbearing potential as determined by medical history and physical examination
* Have body mass indexes of 18 to 35 kilograms per square meter (kg/m^2), inclusive, at screening
* Have screening low density lipoprotein-C (LDL-C) of between 100 and 180 milligrams per deciliter (mg/dL), inclusive, while having taken a stable dose of statin

Exclusion Criteria:

* Have known allergies to compounds related to LY3015014 or any components of the formulation or known clinically significant hypersensitivity to biologic agents
* Have a history of atopy, significant allergies to humanized monoclonal antibodies, clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions [including but not limited to erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis]
* Have significant history of or current cardiovascular (excluding controlled hypertension), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study medication, or of interfering with the interpretation of data
* Have received any vaccine(s) within 1 month of LY3015014 dosing or intend to do so during the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who discontinued from the study prior to completion were permitted to be replaced.
Groups:
- 1.0 mg/kg of LY3015014: LY3015014: 1.0 milligram per kilogram (mg/kg) of LY3015014 subcutaneously (SQ) on 2 dosing occasions occurring 4 weeks apart (Q4W) (Days 1 and 29).
- Placebo: Placebo: 0.9% sodium chloride injection SQ (to match LY3015014) on 2 dosing occasions Q4W (Days 1 and 29).
Period: Overall Study
Arm/Group | 1.0 mg/kg of LY3015014 | Placebo
Started | 11 (1 participant who dropped out was replaced.) | 2
Received at Least 1 Dose of Study Drug | 11 | 2
Completed | 10 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 1.0 mg/kg of LY3015014: LY3015014: 1.0 mg/kg of LY3015014 SQ on 2 dosing occasions (Q4W) (Days 1 and 29).
- Total: Total of all reporting groups
Arm/Group | 1.0 mg/kg of LY3015014 | Placebo | Total
Number analyzed (Participants) | 11 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (6.3) | 52.0 (4.2) | 54.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 12
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 2 | 13
Baseline Low Density Lipoprotein (LDL)-C [Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)] | 134.430 (24.559) | 161.060 (1.372) | 138.527 (24.552)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Other Non-Serious Adverse Events (AEs) or Any Serious AEs (SAEs)
Description: Events deemed to be SAEs by the Investigator as related to study drug administration were collected during the study and 30 days following study drug administration. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion (Day 127)
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- 1.0 mg/kg of LY3015014: LY3015014: 1.0 mg/kg of LY3015014 SQ on 2 dosing occasions Q4W (Days 1 and 29).
Arm/Group | 1.0 mg/kg of LY3015014 | Placebo
Number analyzed (Participants) | 11 | 2
Participants
  AEs | 3 | 1
  SAEs | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3015014
Description: The Cmax was calculated after each dose of LY3015014.
Time Frame: Day 1 and 29: 4 hours (h) and 24 h postdose
Population: Full analysis set (FAS): Data from all randomized participants who received at least 1 dose of the study drug according to the treatment the participants actually received and had evaluable PK data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | 1.0 mg/kg of LY3015014
Number analyzed (Participants) | 11
micrograms per milliliter (µg/mL)
  After Day 1 dosing | 5.06 (36)
  After Day 29 dosing: number analyzed (Participants) | 10
  After Day 29 dosing | 5.57 (58)

3. Secondary Outcome: PK: Area Under the Concentration Curve During One Dosing Interval (AUCt) of LY3015014
Description: The AUCt was calculated after each dose of LY3015014.
Time Frame: Day 1 and 29: 4 h and 24 h postdose
Population: FAS: Data from all randomized participants who received at least 1 dose of study drug according to the treatment the participants actually received and had evaluable PK data for AUCt.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (µg*h/mL)
Arm/Group | 1.0 mg/kg of LY3015014
Number analyzed (Participants) | 10
microgram*hour per milliliter (µg*h/mL)
  After Day 1 dosing | 1960 (37)
  After Day 29 dosing | 2150 (46)

4. Secondary Outcome: PK: Time of Maximum Concentration (Tmax) of LY3015014
Description: tmax was calculated after each dosing of LY3015014 and is reported as the number of days for observed maximum concentration of LY3015014.
Time Frame: Day 1 and 29: 4 h and 24 h postdose
Population: FAS: Data from all randomized participants who received at least 1 dose of study drug according to the treatment the participants actually received and had evaluable PK data for tmax.
Measure: Median (Full Range); unit: days
Arm/Group | 1.0 mg/kg of LY3015014
Number analyzed (Participants) | 11
days
  After Day 1 dosing | 4 [4 to 4]
  After Day 29 dosing: number analyzed (Participants) | 10
  After Day 29 dosing | 5 [5 to 5]

5. Secondary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percentage change from baseline in LDL-C was calculated as Least Squares (LS) mean using mixed model repeated measures (MMRM) analysis adjusted for baseline measurement. Treatment, day after dosing, and treatment-by-day interaction were included in the model.
Time Frame: Baseline, Day 43 and Day 57
Population: Pharmacodynamic analyses set: Participants who received at least 1 dose of investigational product according to the treatment actually received and had a baseline measurement and at least 1 post baseline measurement for LDL-C.
Measure: Least Squares Mean (90% Confidence Interval); unit: µg/mL
Groups:
- Placebo: Placebo: 0.9% sodium chloride injection given SQ (to match LY3015014) on 2 dosing occasions Q4W (Days 1 and 29).
Arm/Group | 1.0 mg/kg of LY3015014 | Placebo
Number analyzed (Participants) | 11 | 2
µg/mL
  Day 43 | -49.10 [-57.34 to -40.87] | 1.38 [-17.51 to 20.27]
  Day 57 | -37.53 [-45.79 to -29.27] | 7.58 [-11.31 to 26.47]
Statistical Analysis 1: Comparison: 1.0 mg/kg of LY3015014 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis — P-value is for Day 43; Mean Difference (Net) = -50.49, 90% CI 2-sided [-71.27 to -29.70]
Statistical Analysis 2: Comparison: 1.0 mg/kg of LY3015014 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Effects Models Analysis — P-value is for Day 57; Mean Difference (Net) = -45.11, 90% CI 2-sided [-65.91 to -24.31]

ADVERSE EVENTS:
Time Frame: Baseline through Study Completion (Day 127)
Arm/Group | 1.0 mg/kg of LY3015014 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/2
Other Adverse Events (participants affected / at risk) | 3/11 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0 mg/kg of LY3015014 (N=11) | Placebo (N=2)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days